CLINICAL TRIAL: NCT02048436
Title: Perminova Respiratory Effort Accuracy Validation 09-12-2013-Rev 2
Status: Completed | Type: Observational
Sponsor: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 78o944o
Record Dates: First submitted 2013-09-25; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Respiratory Rate Accuracy Test
Keywords: Respiratory Rate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- male female 18-45 years range of body types: 18 male female subject mix that are 18-45 years of age and selected to represent a range of body types of varying physiques and body mass indexes

SUMMARY:
The purpose of this study is to validate the accuracy of the Perminova N4 Monitoring system Respiration Rate technology.

DETAILED DESCRIPTION:
After IRB Approval, eighteen volunteer test subjects will be entered into an accuracy study that is designed to validate accuracy of the respiratory rate technology of the Perminova N4 Monitoring system (Device Under Test). The subjects will be selected to represent a range of body types including small, average, muscular, and large with a range of BMI's.

A range of stable respiratory rates will be elicited from each volunteer test subject. The rates will be approximately 5, 10, 15, 20, 25, 30, 35 and 40 breaths per minute; with some natural variation from these exact numbers.

Each subject will be instrumented with an open system mask that allows for measurement of the end tidal carbon dioxide (EtCO2) respiratory rate and tidal volume. The EtCO2 monitor will be used as the Accuracy Reference Device (Reference) in this study. Performance of the currently released ECG Impedance Respiratory Rate monitor (Acceptance Standard) will be used to establish the acceptance criteria in this study by comparing to Reference.

ELIGIBILITY:
Inclusion Criteria:

* male
* female
* 18-45
* range of physiques
* healthy

Exclusion Criteria:

* injury to sensor area
* skin inflammation
* implanted devices such as pacemakers
* pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy Male or female, ages 18-45
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate of test subject as compared to end tidal CO2 | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark Laboratory, Louisville, Colorado, United States